CLINICAL TRIAL: NCT04562740
Title: ABLUMINUS Below the Knee (BTK) Drug Eluting Stent (DES) Registry (ABLUMINUS BTK) - First in Men
Brief Title: ABLUMINUS DES BTK Registry - FIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLUMINUS BTK
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Artery Disease; Arterial Disease of Legs; Atherosclerosis
Keywords: Sirolimus; DES; PAD; PTA
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: During the index angioplasty revascularisation procedure of the limb salvage programme, the ABLUMINUS DES drug eluting stent will be deployed after successful conventional balloon angioplasty.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABLUMINUS DES (Experimental): ABLUMINUS DES drug eluting stent will be deployed after successful conventional balloon angioplasty.
  Sirolimus drug dosage on the ABLUMINUS DES drug eluting stent system is determined by Concept Medical to deliver the optimal dose of sirolimus to the abluminal surface of the BTK lesions.
  Interventions: Device: ABLUMINUS DES drug eluting stent

INTERVENTIONS:
Device: ABLUMINUS DES drug eluting stent — Following successful plain balloon angioplasty of the arterial lesion, (defined as <30% residual stenosis after treatment at rated burst pressure of the angioplasty balloon), the ABLUMINUS stent will be deployed at the lesion as per Instructions for Use (IFU) after appropriate sizing using the diameter of the plain balloon angioplasty. After deployment of the ABLUMINUS stent, further balloon angioplasty of the stent will be performed, using the same diameter standard balloon catheter at 2 minutes inflation, to ensure adequate moulding and expansion of the stent.

SUMMARY:
A prospective, single center, single arm non-randomized trial collecting safety and effectiveness data for the ABLUMINUS DES System to treat BTK lesions in subjects with CLI.

DETAILED DESCRIPTION:
The burden of limb loss as a result of peripheral arterial disease (PAD) is high and this problem is set to worsen globally with increasing prevalence of diabetes. Treatment of PAD in diabetic critical limb ischemia (CLI) primarily involves revascularisation of the limb. Angioplasty as a first line strategy of revascularization over surgical procedures has been adopted by most vascular centers.

Arterial blockages for diabetic CLI patients occur predominantly in below the knee arteries which can be challenging to treat effectively. This is due to the high incidence of arterial recoil after conventional balloon angioplasty due the natural tendency of the vessels to maintain their original shape and the high restenosis rates of calcified lesions.

To address these problems the novel ABLUMINUS DES system is specifically designed to withstand the mechanical recoil of diseased BTK arteries whilst delivering sirolimus to biologically inhibit restenosis.

This study postulates that the application of the ABLUMINUS DES system will be safe and will result in better vascular patency in BTK arteries for CLI patients.

The investigators aim to conduct a prospective, all comers, single arm, single centre registry of the ABLUMINUS DES system for the treatment of BTK disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 21 years or older and has signed and dated the trial informed consent document (ICD)
2. Subject is willing and able to comply with the trial testing, procedures and follow-up schedule
3. Subject has chronic, symptomatic diabetic related lower limb ischemia, determined by Rutherford categories 4 to 6 in the target limb, with wound(s) confined to toes/forefoot
4. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active must be using, or agree to use, a medically-acceptable method of birth control as confirmed by the investigator

Intraoperative inclusion criteria

1. Occlusive target lesion(s) located in the tibioperoneal trunk, anterior tibial, posterior tibial and/or peroneal artery(ies).
2. Target lesion(s) must be at least 4cm above the ankle joint
3. Degree of stenosis ≥ 70% by visual angiographic assessment
4. RVD is between 2.5 - 3.75mm
5. Total target lesion length (or series of lesion segments) to be treated is > 200 mm
6. Target lesion(s) is located in an area that may be stented without blocking access to patent main branches
7. Treatment of all above the knee inflow lesion(s) is successful prior to treatment of the target lesion
8. Guidewire has successfully crossed the target lesion(s)

Exclusion Criteria:

1. Life expectancy ≤ 1year
2. Stroke ≤ 90 days prior to the procedure date
3. Prior or planned major amputation in the target limb
4. Previous surgery in the target vessel(s) (including prior ipsilateral crural bypass)
5. Previously implanted stent in the target vessel(s)
6. Failed PTA of target lesion/vessel ≤ 60 days prior to the procedure date
7. Heel gangrene
8. Subject has a platelet count ≤ 50 or ≥ 600 X 103/µL ≤ 30 days prior to the procedure date
9. NYHA class IV heart failure
10. Subject has symptomatic coronary artery disease (ie, unstable angina)
11. History of myocardial infarction or thrombolysis ≤ 90 days prior to the procedure date
12. Non-atherosclerotic disease resulting in occlusion (eg, embolism, Buerger's disease, vasculitis)
13. Subject is currently taking Canagliflozin
14. Body Mass Index (BMI) <18
15. Active septicemia or bacteremia
16. Coagulation disorder, including hypercoagulability
17. Contraindication to anticoagulation or antiplatelet therapy
18. Known allergies to stent or stent components
19. Known allergy to contrast media that cannot be adequately pre-medicated prior to the interventional procedure
20. Known hypersensitivity to heparin
21. Subject is on a high dose of steroids or is on immunosuppressive therapy
22. Subject is currently participating, or plans to participate in, another investigational trial that may confound the results of this trial (unless written approval is received from the Concept Medical study team)

Intraoperative exclusion criteria

1. Angiographic evidence of intra-arterial acute/subacute thrombus or presence of atheroembolism
2. Treatment required in > 2 target vessels (Note: a target lesion originating in one vessel and extending into another vessel is considered 1 target vessel)
3. Treatment requires the use of alternate therapy in the target vessel(s)/lesion(s), (eg, atherectomy, cutting balloon, re-entry devices, laser, radiation therapy)
4. Aneurysm is present in the target vessel(s)
5. Extremely calcified lesions
6. Failure to obtain <30% residual stenosis in a pre-existing lesion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Primary patency using duplex ultrasound at 6 months post-procedure | at 6 months post-procedure
  Number of Primary patency using duplex ultrasound at 6 months post-procedure
Major adverse events (MAE) at 6 months post-procedure | at 6 months post-procedure
  Number of Major adverse events (MAE) (MAE is defined as above ankle amputation in index limb; major re-intervention; and perioperative (30 day) mortality)

SECONDARY OUTCOMES:
Primary and assisted primary patency | 6, 12, 24 months post procedure
  Target lesion patency rate measured by duplex ultrasound
Clinically driven target lesion revascularization | 1, 3, 6, 12, 24 months post procedure
  Number of Clinically-driven target lesion revascularization
Major amputation rates | 1, 3, 6, 12, 24 months post procedure
  Rates of amputation of the lower limb at the ankle level or above
Subject quality-of-life values by change in EQ-5D (EuroQol 5 dimension) | 1, 3, 6 and 12 months post procedure
  The EQ-5D is a descriptive system of health-related quality-of-life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 5 responses. The responses record 5 levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension). The levels are assigned a numeric code 1-5 (eg, 1= no problems and 5= extreme problems). Sub-scores are not applicable.
Wound Assessment | 1, 3, 6, 12, 24 months post procedure
  Descriptive characteristics of wound healing will be recorded
Rutherford classification | 3, 6, 12, 24 months post procedure
  Change in Rutherford classification as assessed by the investigator
Adverse Events | 1, 3, 6, 12, 24 months post procedure
  Number of Adverse events
Unplanned hospital readmission | Up to 30 days post procedure
  Unplanned hospital related to Critical Limb Ischemia readmission rate
All Cause Mortality | 6, 12, 24 months years post procedure
  Number of patients with all-cause death
Hemodynamic outcomes | 6 and 12 months post procedure
  Changes in ankle brachial index (ABI) and/or Toe pressures (TP

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Romiti M, Albers M, Brochado-Neto FC, Durazzo AE, Pereira CA, De Luccia N. Meta-analysis of infrapopliteal angioplasty for chronic critical limb ischemia. J Vasc Surg. 2008 May;47(5):975-981. doi: 10.1016/j.jvs.2008.01.005. Epub 2008 Apr 18. PMID 18372148
- [Background] Siablis D, Karnabatidis D, Katsanos K, Diamantopoulos A, Spiliopoulos S, Kagadis GC, Tsolakis J. Infrapopliteal application of sirolimus-eluting versus bare metal stents for critical limb ischemia: analysis of long-term angiographic and clinical outcome. J Vasc Interv Radiol. 2009 Sep;20(9):1141-50. doi: 10.1016/j.jvir.2009.05.031. Epub 2009 Jul 19. PMID 19620014
- [Background] Biondi-Zoccai GG, Sangiorgi G, Lotrionte M, Feiring A, Commeau P, Fusaro M, Agostoni P, Bosiers M, Peregrin J, Rosales O, Cotroneo AR, Rand T, Sheiban I. Infragenicular stent implantation for below-the-knee atherosclerotic disease: clinical evidence from an international collaborative meta-analysis on 640 patients. J Endovasc Ther. 2009 Jun;16(3):251-60. doi: 10.1583/09-2691.1. PMID 19642789
- [Background] Kudo T, Chandra FA, Ahn SS. The effectiveness of percutaneous transluminal angioplasty for the treatment of critical limb ischemia: a 10-year experience. J Vasc Surg. 2005 Mar;41(3):423-35; discussion 435. doi: 10.1016/j.jvs.2004.11.041. PMID 15838475
- [Background] Scheinert D, Katsanos K, Zeller T, Koppensteiner R, Commeau P, Bosiers M, Krankenberg H, Baumgartner I, Siablis D, Lammer J, Van Ransbeeck M, Qureshi AC, Stoll HP; ACHILLES Investigators. A prospective randomized multicenter comparison of balloon angioplasty and infrapopliteal stenting with the sirolimus-eluting stent in patients with ischemic peripheral arterial disease: 1-year results from the ACHILLES trial. J Am Coll Cardiol. 2012 Dec 4;60(22):2290-5. doi: 10.1016/j.jacc.2012.08.989. PMID 23194941
- [Background] Bosiers M, Scheinert D, Peeters P, Torsello G, Zeller T, Deloose K, Schmidt A, Tessarek J, Vinck E, Schwartz LB. Randomized comparison of everolimus-eluting versus bare-metal stents in patients with critical limb ischemia and infrapopliteal arterial occlusive disease. J Vasc Surg. 2012 Feb;55(2):390-8. doi: 10.1016/j.jvs.2011.07.099. Epub 2011 Dec 14. PMID 22169682
- [Background] Rastan A, Tepe G, Krankenberg H, Zahorsky R, Beschorner U, Noory E, Sixt S, Schwarz T, Brechtel K, Bohme C, Neumann FJ, Zeller T. Sirolimus-eluting stents vs. bare-metal stents for treatment of focal lesions in infrapopliteal arteries: a double-blind, multi-centre, randomized clinical trial. Eur Heart J. 2011 Sep;32(18):2274-81. doi: 10.1093/eurheartj/ehr144. Epub 2011 May 26. PMID 21622669